CLINICAL TRIAL: NCT05097326
Title: Mifepristone as an Adjunct to Transcervical Balloon for Labor Induction (MiLI): A Randomized Clinical Trial
Brief Title: Mifepristone for Labor Induction
Acronym: MiLI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 62448
Record Dates: First submitted 2021-10-15; First posted 2021-10-28 (Actual); Results first posted 2024-07-31 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Induced Vaginal Delivery
MeSH Terms: interventions — Mifepristone; Misoprostol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mifepristone (Active Comparator): Participants will be given mifepristone with insertion of the cervical Cook balloon for labor induction
  Interventions: Drug: Mifepristone
- Misoprostol (Active Comparator): Participants will be given misoprostol with insertion of the cervical Cook balloon for labor induction
  Interventions: Drug: Misoprostol

INTERVENTIONS:
Drug: Mifepristone — Mifepristone 200mg taken orally
  Arms: Mifepristone
Drug: Misoprostol — Misoprostol 50 mcg taken orally, and may receive additional doses of misoprostol 50 - 100 mcg as needed
  Arms: Misoprostol

SUMMARY:
The purpose of this trial is to explore mifepristone as an option for induction of labor at term by evaluating the efficacy of mifepristone use for cervical preparation. Since the Labor Induction versus Expectant Management in Low-Risk Nulliparous Women (ARRIVE) trial supporting that elective induction after 39 weeks decreases cesarean sections and morbidity, rates of elective term inductions are increasing.

At Lucile Packard Children's Hospital at Stanford University specifically, approximately 40% of spontaneous vaginal deliveries follow induction of labor, with an average induction time of 20 hours. Previous studies have established the maternal and neonatal safety of mifepristone in term inductions, however, this study will assess the difference in overall time from induction to complete cervical dilation, delivery, and the total time on Labor and Delivery.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant patients between ages 18 to 45 years
2. Singleton, live gestation
3. Nulliparous
4. Gestational age between 37 weeks 0 days - 42 weeks 0 days
5. Fetus in cephalic presentation
6. Patients admitted for labor induction
7. Patients who are not in labor with intact membranes
8. Patients with no contraindication for vaginal delivery (placenta previa, vasa previa, active genital herpes)
9. Patients with no contraindications for mifepristone (chronic adrenal failure, concurrent long-term corticosteroid therapy, history of allergy to mifepristone, or other prostaglandins, hemorrhagic disorders or concurrent anticoagulant therapy, inherited porphyria, or an intrauterine device (IUD) in place)
10. Patients with a Bishop score <6 at time of randomization
11. Transcervical balloon in place <3 hours prior to the time of randomization without prior cervical preparation

Exclusion Criteria:

1. Significant cardiac, renal, or hepatic maternal comorbidities, severe gestational hypertension or preeclampsia with severe features
2. Pregnancies complicated by major fetal anomalies
3. Patients with a uterine scar
4. Pregnancies complicated by fetal growth restriction (Estimated fetal weight <10%)
5. Pregnancies complicated by oligohydramnios
6. Fetuses with an estimated fetal weight >4500 gm by recent ultrasound or Leopold's exam on admission
7. Patients with class 3 obesity (BMI >40)
8. Fetuses with a persistent category 2 or 3 fetal heart tracing at labor induction admission
9. Vaginal bleeding at the time of randomization
10. Any indication for scheduled cesarean delivery
11. Hypersensitivity to oxytocin
12. Uterine contractions equal to or greater than 5 in 10 minutes for sustained 30 minutes
13. Hypersensitivity to prostaglandins

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-06-27 (Actual); Primary Completion 2023-04-29 (Actual); Study Completion 2023-04-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Lucile Packard Children's Hospital, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Mifepristone: Mifepristone 200 mg orally plus cervical Cook balloon
- Misoprostol: Misoprostol 50 mcg orally plus cervical Cook balloon
Period: Overall Study
Arm/Group | Mifepristone | Misoprostol
Started | 15 | 15
Received Medication | 14 | 15
Completed | 14 | 15
Not Completed | 1 | 0
Not completed — Spontaneous labor prior to medication administration | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mifepristone | Misoprostol | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.46 (4.64) | 31.21 (7.07) | 30.82 (5.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 15 | 30
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 7 | 17
  Not Hispanic or Latino | 4 | 8 | 12
  Unknown or Not Reported | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 4 | 4 | 8
  White | 2 | 5 | 7
  Other | 8 | 6 | 14
  Unknown | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Uterine Contractions
Description: Measured total number of uterine contractions per hour - with and without fetal heart rate decelerations.
Time Frame: Up to approximately 72 hours, from start of labor induction to removal of transcervical balloon
Population: Intent to treat analysis set: all participants who were randomized regardless of what treatment (if any) they received.
Measure: Median (Inter-Quartile Range); unit: contractions
Arm/Group | Mifepristone | Misoprostol
Number analyzed (Participants) | 15 | 15
contractions
  Total | 103 [68 to 156] | 112 [84 to 186]
  Per hour | 9 [6 to 13] | 15 [9 to 17]
Statistical Analysis 1: Comparison: Mifepristone vs Misoprostol; Analysis of total contractions; Test type: Other; p = 0.44, Fisher Exact — a p-value <0.05 would be considered statistically significant
Statistical Analysis 2: Comparison: Mifepristone vs Misoprostol; Analysis of contractions per hour; Test type: Other; p = 0.02, Fisher Exact — a p-value of <0.05 would be considered statistically significant

2. Primary Outcome: Number of Participants With Uterine Tachysystole
Description: Participants with uterine tachysystole (more than 5 contractions in 10 minutes with and without fetal heart rate decelerations) .
Time Frame: Up to approximately 72 hours from start of labor induction
Population: Intent to treat analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Mifepristone | Misoprostol
Number analyzed (Participants) | 15 | 15
Participants
  Uterine tachysystole-12 hours post administration | 0 | 5
  Uterine tachysystole- total labor duration | 1 | 5
Statistical Analysis 1: Comparison: Mifepristone vs Misoprostol; Comparison at 12 hours after labor induction; Test type: Other; p = 0.04, Fisher Exact — a p-value of <0.05 would be considered statistically significant
Statistical Analysis 2: Comparison: Mifepristone vs Misoprostol; Comparison of uterine tachysystole of total labor duration; Test type: Other; p = 0.17, Fisher Exact — a p-value of <0.05 would be considered statistically significant

3. Primary Outcome: Number of Minutes in Hypertonus
Description: Time in hypertonus (a single contraction lasting more than 2 minutes) per hour.
Time Frame: Up to approximately 72 hours, from start of labor induction until the time of delivery
Population: Intent to treat analysis set
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Mifepristone | Misoprostol
Number analyzed (Participants) | 15 | 15
minutes | 1.33 (5.16) | 0.93 (2.49)
Statistical Analysis 1: Comparison: Mifepristone vs Misoprostol; Test type: Other; p = 0.63, Wilcoxon (Mann-Whitney) — a p-value <0.05 would be considered statistically significant

4. Primary Outcome: Time to Complete Cervical Dilation
Description: Total time from start of labor induction to complete cervical dilation (10 cm).
Time Frame: Up to approximately 72 hours from start of labor induction
Population: Intent to treat analysis set
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Mifepristone | Misoprostol
Number analyzed (Participants) | 15 | 15
hours | 24.0 [16.0 to 33.0] | 16.0 [11.0 to 22.0]
Statistical Analysis 1: Comparison: Mifepristone vs Misoprostol; Test type: Other; p = 0.01, Wilcoxon (Mann-Whitney) — a p-value of <0.05 would be considered statistically significant

5. Primary Outcome: Time to Delivery
Time Frame: Up to approximately 72 hours, from start of labor induction until the time of delivery
Population: Intent to treat analysis set
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Mifepristone | Misoprostol
Number analyzed (Participants) | 15 | 15
hours | 26.0 [12.0 to 39.0] | 19.0 [13.0 to 26.0]
Statistical Analysis 1: Comparison: Mifepristone vs Misoprostol; Comparison at complete cervical dilation; Test type: Other; p = 0.04, Wilcoxon (Mann-Whitney) — a p-value of <0.05 would be considered statistically significant

6. Primary Outcome: Total Labor and Delivery Unit Admission Duration Time
Description: Total time on Labor & Delivery from the time of admission to the time of transfer to postpartum unit
Time Frame: Up to approximately 80 hours after the time of Labor and delivery admission
Population: Intent to treat analysis set
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Mifepristone | Misoprostol
Number analyzed (Participants) | 15 | 15
hours | 29.0 [24.0 to 41.0] | 21.0 [15.0 to 32.0]
Statistical Analysis 1: Comparison: Mifepristone vs Misoprostol; Comparison at postpartum transfer; Test type: Other; p = 0.04, Wilcoxon (Mann-Whitney) — a p-value of <0.05 would be considered statistically significant

7. Primary Outcome: Number of Patients Who Undergo Cesarean Delivery
Time Frame: Up to approximately 72 hours from start of labor induction
Population: Intent to treat analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Mifepristone | Misoprostol
Number analyzed (Participants) | 15 | 15
Participants | 5 | 2
Statistical Analysis 1: Comparison: Mifepristone vs Misoprostol; Test type: Other; p = 0.68, Fisher Exact — a p-value of <0.05 would be considered statistically significant

8. Primary Outcome: Number of Patients Able to Achieve Active Labor
Description: Active labor defined as cervical of dilation >=6 cm.
Time Frame: Up to approximately 72 hours from start of labor induction
Population: Intent to treat analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | Mifepristone | Misoprostol
Number analyzed (Participants) | 15 | 15
Participants | 13 | 13
Statistical Analysis 1: Comparison: Mifepristone vs Misoprostol; Test type: Other; p = 1, Fisher Exact — A p-value of <0.05 would be considered significant

9. Primary Outcome: Number of Patients With Severe Maternal Morbidity
Description: Number of participants with serious maternal morbidity based on CDC criteria for major maternal morbidity and mortality
Time Frame: Up to approximately 1 week after hospital admission for delivery
Population: Intent to treat analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Mifepristone | Misoprostol
Number analyzed (Participants) | 15 | 15
Participants | 0 | 1
Statistical Analysis 1: Comparison: Mifepristone vs Misoprostol; Test type: Other; p = 1, Fisher Exact — a p-value of <0.05 would be considered statistically significant

10. Primary Outcome: Mean Neonatal Arterial Cord Blood pH
Description: Laboratory values for neonatal arterial cord blood pH. Arterial pH lower than 7.0 indicates metabolic acidosis.
Time Frame: Within approximately 2 hours after delivery (approximately 5 minutes to obtain sample)
Population: Neonatal cords available for analysis
Measure: Mean (Standard Deviation); unit: pH
Units Other Than Participants: Neonatal cords
Arm/Group | Mifepristone | Misoprostol
Number analyzed (Participants) | 12 | 11
Number analyzed (Neonatal cords) | 12 | 11
pH | 7.16 (0.06) | 7.17 (0.06)
Statistical Analysis 1: Comparison: Mifepristone vs Misoprostol; Test type: Other; p = 0.90, Wilcoxon (Mann-Whitney) — A p-value <0.05 would be considered statistically significant

11. Primary Outcome: Number of Participants With Neonatal APGAR Score <7
Description: Compare the APGAR scores (at 1 and 5 minutes). The Apgar score comprises five components: 1) color, 2) heart rate, 3) reflexes, 4) muscle tone, and 5) respiration, each of which is given a score of 0, 1, or 2; scores are summed for an overall score of 0 to 10 (higher scores reflect better neonatal outcomes).
Time Frame: At 1 minute and 5 minutes of infant life (approximately 10 seconds to perform each assessment)
Population: Neonates are included in the analysis but were not considered enrolled in the study.
Measure: Count of Units; unit: Neonates
Units Other Than Participants: Neonates
Arm/Group | Mifepristone | Misoprostol
Number analyzed (Participants) | 15 | 15
Number analyzed (Neonates) | 15 | 15
Neonates
  1 minute | 5 | 1
  5 minutes | 1 | 0
Statistical Analysis 1: Comparison: Mifepristone vs Misoprostol; 1 minute APGAR score; Test type: Other; p = 0.17, Fisher Exact — a p-value <0.05 would be considered statistically significant
Statistical Analysis 2: Comparison: Mifepristone vs Misoprostol; APGAR score at 5 minutes; Test type: Other; p = 1, Fisher Exact — A p-value of <0.05 would be statistically significant

12. Primary Outcome: Number of Patients With Serious Neonatal Morbidity
Description: Defined as need for respiratory support within 72 hours after birth, hypoxic-ischemic encephalopathy, seizure, infection, meconium aspiration syndrome, intracranial or subgaleal hemorrhage, hypotension requiring vasopressor support, admission to neonatal intensive care unit
Time Frame: Up to 7 days after birth
Population: Neonates are included in the analysis but were not considered enrolled in the study.
Measure: Count of Units; unit: Neonates
Units Other Than Participants: Neonates
Arm/Group | Mifepristone | Misoprostol
Number analyzed (Participants) | 15 | 15
Number analyzed (Neonates) | 15 | 15
Neonates | 3 | 0
Statistical Analysis 1: Comparison: Mifepristone vs Misoprostol; Test type: Other; p = 0.22, Fisher Exact — A p-value of <0.05 would be considered statistically significant

ADVERSE EVENTS:
Time Frame: Average approximately 2 to 3 days.
Arm/Group | Mifepristone | Misoprostol
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 3/15 | 1/15
Other Adverse Events (participants affected / at risk) | 1/15 | 0/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mifepristone (N=15) | Misoprostol (N=15)
Unanticipated NICU admission (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Hysterectomy, postpartum hemorrhage (Pregnancy, puerperium and perinatal conditions) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mifepristone (N=15) | Misoprostol (N=15)
5 min APGAR <7 (Pregnancy, puerperium and perinatal conditions) | 1 | 0 — Not related

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-11): https://cdn.clinicaltrials.gov/large-docs/26/NCT05097326/Prot_SAP_000.pdf